CLINICAL TRIAL: NCT03859479
Title: A Prospective Randomized Controlled Trial of Cold Snare Polypectomy vs. Conventional Polypectomy for Non-pedunculated Colorectal Adenomas
Brief Title: Cold Snare Polypectomy of Non-pedunculated Colorectal Adenomas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 122
Record Dates: First submitted 2019-02-28; First posted 2019-03-01 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Colorectal Polyp
Keywords: Cold snare polypectomy; Hot snare polypectomy; Сolorectal polyps; Endoscopic treatment

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold snare polypectomy (Experimental): After a target polyp was identified, it should be placed at the comfortable position. Then the snare will be opened and encircled the polyp without air aspiration. Then, the snare will be captured the polyp with at least 1-2 mm of surrounding normal tissue. The polyp will be guillotined and would not be lifted or tented until complete closure is achieved. After resection, the mucosal defect the marginal mucosa was carefully observed, with used of magnification and image enhancement. If residual polyp tissue was recognised, additional removal using the cold snare technique or biopsy forceps will be performed. If a submucosal injection prior to snaring was necessary it will be permitted. After polypectomy all patients will be observed for 3-4 days in-hospital
  Interventions: Procedure: Cold snare polypectomy
- Hot snare polypectomy (Active Comparator): After a target polyp was identified, it should be placed at the comfortable position. Then the polyp with minimal normal tissue will be captured by the snare. The ensnared polyp should be tented away from the colonic wall and removed by one the types of electric currents. After resection, the mucosal defect will be washed thoroughly and the marginal mucosa was carefully observed, with used of magnification and image enhancement, such as near focus imaging or narrow band imaging. If a submucosal injection prior to snaring was necessary it would be permitted. If residual polyp tissue was recognised, additional removal using coagulation or biopsy forceps will be performed. After polypectomy all patients will be observed for 3-4 days in-hospital
  Interventions: Procedure: Hot snare polypectomy

INTERVENTIONS:
Procedure: Cold snare polypectomy — After a target polyp was identified, it should be placed at the comfortable position. Then the snare will be opened and encircled the polyp without air aspiration. Then, the snare will be captured the polyp with at least 1-2 mm of surrounding normal tissue. The polyp will be guillotined and would not be lifted or tented until complete closure is achieved. After resection, the mucosal defect the marginal mucosa was carefully observed, with used of magnification and image enhancement. If residual polyp tissue was recognised, additional removal using the cold snare technique or biopsy forceps will be performed. If a submucosal injection prior to snaring was necessary it will be permitted. After polypectomy all patients will be observed for 3-4 days in-hospital
  Arms: Cold snare polypectomy
Procedure: Hot snare polypectomy — After a target polyp was identified, it should be placed at the comfortable position. Then the polyp with minimal normal tissue will be captured by the snare. The ensnared polyp should be tented away from the colonic wall and removed by one the types of electric currents. After resection, the mucosal defect will be washed thoroughly and the marginal mucosa was carefully observed, with used of magnification and image enhancement, such as near focus imaging or narrow band imaging. If a submucosal injection prior to snaring was necessary it would be permitted. If residual polyp tissue was recognised, additional removal using coagulation or biopsy forceps will be performed. After polypectomy all patients will be observed for 3-4 days in-hospital
  Arms: Hot snare polypectomy

SUMMARY:
A prospective randomised controlled trial of cold vs hot snare polypectomy of non-pedunculated colorectal adenomas.

DETAILED DESCRIPTION:
Diagnostic colonoscopy will be performed in all patients. If a polyp, appropriate for inclusion criteria, is identified, an endoscopic polypectomy will be assigned. All eligible polyps will be randomly assigned (1:1) to endoscopic polypectomy with either the cold snare resection or hot snare resection (control group). Randomization will be stratified using random numbers. After resection, the marginal mucosa will be carefully observed with used of magnification and image enhancement (near focus imaging or narrow band imaging) for determine residual tissue. The time period when the snare will be entered in the bowel lumen and until a polyp will be retrieved will be recorded by a stopwatch.

All polyps will be retrieved for morphological examination to estimate R0/R1resetion. After polypectomy all patients will be observed for 3-4 days in-hospital to diagnose and eliminate complications (delayed bleeding and perforations). All patients will have a control colonoscopy 6 months after polypectomy to investigate long-term results.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-pedunculated colorectal adenomas who had provided written informed consent

Exclusion Criteria:

* known coagulopathy.
* polyposis of the alimentary tract.
* inflammatory bowel disease.
* malignant polyps.
* associated diseases in the stage of decompensation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-01-20 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 14 days
Complete resection rate | 1 day

SECONDARY OUTCOMES:
Incidence of local recurrence | 6 months
The immediate bleeding or immediate perforation rate after polypectomy | 1 day
Complication rate | 14 days
Use of submucosal injection | 1 day
Polyp retrieval rate | 1 day
The procedure time | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- State Scientific Centre of Coloproctology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No